CLINICAL TRIAL: NCT02295293
Title: The Effects of Rhus Coriaria L. (Rhus or Somagh) on Serum Lipid Levels of Patients With Hyperlipidemia
Brief Title: The Effects of Rhus Coriaria L. on Serum Lipid Levels of Patients With Hyperlipidemia
Acronym: SomaghLipid
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mesbah Shams, MD, Associate professor of Internal Medicine & Endocrinology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P-92-5581
Record Dates: First submitted 2014-11-10; First posted 2014-11-20 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Hyperlipidemias
Keywords: Rhus; Cholesterol; Triglycerides; Lipids; Medicine, Traditional; Herbal medicine
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rhus (Experimental): 500 mg of Rhus Coriaria L. (Rhus) powder in capsule: 1 capsule twice daily for 6 weeks
  Interventions: Drug: Rhus Coriaria L. (Rhus)
- Placebo (Placebo Comparator): Placebo capsule: 1 capsule twice daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rhus Coriaria L. (Rhus) — 500 mg of Rhus Coriaria L. (Rhus) powder in capsule: 1 capsule twice daily for 6 weeks
  Arms: Rhus
Drug: Placebo — Placebo capsule: 1 capsule twice daily for 6 weeks
  Arms: Placebo

SUMMARY:
Coronary heart disease and stroke are two main causes of human deaths and is directly related to increased levels of plasma lipids.High total cholesterol and low high density lipoprotein cholesterol concentrations are often associated with endothelium dysfunction and inflammation, which can be followed by atherosclerosis.

Rhus coriaria L. (Rhus) with the public name of "Somagh" is a plant species in the anacardiaceae family that is used as a food supplement, spice in Middle East region (Iran, Turkey and Arabic countries).

In a double blind randomized placebo-controlled clinical trial, the investigators want to evaluate the effects of Somagh (Rhus coriaria L.) on serum lipid levels of patients with hyperlipidemia.

DETAILED DESCRIPTION:
Rhus (Somagh) is found in temperate and tropical regions worldwide, often growing in areas of marginal agricultural capacity. Rhus is used as an herbal remedy in traditional medicine because of its assumed analgesic, antidiarrhetic, antiseptic, anorexic and antihypergylcemic properties. The fruits of Rhus contain flavonols, phenolic acids, hydrolysable tannins, anthocyans and organic acids such as malice, citric and tartaric acids. Some studies have shown that polyphenols could have beneficial effects on cardiovascular disease and cancer and could be regarded as bioactive compounds with a high potential health-promoting capacity. Phenolic compounds inhibit lipid peroxidation, scavenge the superoxide anion and hydroxyl radical, and enhance the activities of detoxifying enzymes.Moreover, the hypocholesterolemic action of dietary polyphenols has been reported. The hypocholesterolemic effect of Rhus fruit powder and its components have been reported previously in rabbits and mice.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-65 years
* Serum triglyceride >150mg/dl AND/OR total cholesterol >= 240mg/dl

Exclusion Criteria:

* Serum triglyceride > 500 mg/dl
* Serum LDL-cholesterol at level which need drug treatment according to the patient risk categories (NCEP-ATP III)
* Diabetes mellitus
* Hypo. or hyperthyroidism
* Any systemic illnesses e.g. liver cirrhosis, acute or chronic renal failure, heart failure
* Use of drugs: OCPs, lipid lowering agents, thiazides
* Pregnancy
* Alcoholism
* History of allergic reaction to Somagh

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Serum total cholesterol level | 6 weeks
Serum triglyceride level | 6 weeks
Serum HDL-cholesterol level | 6 weeks

SECONDARY OUTCOMES:
Serum LDL-cholesterol level | 6 weeks
Fasting Blood Sugar (FBS) | 6 weeks
Serum creatinin level | 6 weeks
Serum ALT level | 6 weeks
Serum AST level | 6 weeks
Serum alkaline phosphatase level | 6 weeks
Number of patients with adverse events | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mesbah Shams, M.D., Study Chair — Endocrine and Metabolism Research Center, Shiraz University of Medical Sciences, Shiraz, Iran; Majid Nimruzi, M.D., Principal Investigator — Research Center for Traditional Medicine & History of Medicine, Shiraz University of Medical Sciences, Shiraz, Iran; Pooya Faridi, PhD, Principal Investigator — Research Center for Traditional Medicine & History of Medicine, Shiraz University of Medical Sciences, Shiraz, Iran; Mojtaba Heydari, MD, Principal Investigator — Research Center for Traditional Medicine & History of Medicine, Shiraz University of Medical Sciences, Shiraz, Iran
Locations (1):
- Shahid Motahhari Clinic, Shiraz University of Medical Sciences, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Hajmohammadi Z, Heydari M, Nimrouzi M, Faridi P, Zibaeenezhad MJ, Omrani GR, Shams M. Rhus coriaria L. increases serum apolipoprotein-A1 and high-density lipoprotein cholesterol levels: a double-blind placebo-controlled randomized clinical trial. J Integr Med. 2018 Jan;16(1):45-50. doi: 10.1016/j.joim.2017.12.007. Epub 2017 Dec 14. PMID 29397092